CLINICAL TRIAL: NCT02062749
Title: A Phase I Trial With Escalating Doses of Oxaliplatin and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Children and Adolescents With Extensive Colon Carcinoma
Brief Title: Escalating Doses of Oxaliplatin and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Children and Adolescents With Extensive Colon Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0438; NCI-2014-01239 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Colon Cancer; Pediatric; Adolescent; Hyperthermic Intraperitoneal Chemotherapy; HIPEC; Oxaliplatin; Eloxatin
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyperthermic Intraperitoneal Chemotherapy (Experimental): After cytoreductive surgery and lysis of adhesions, two large bore catheters are placed in the peritoneal cavity through the incision. Thirty minutes before HIPEC is begun, body temperature is cooled to 35°C. ). The catheters are connected to a perfusion circuit. Heated Oxaliplatin is added to the perfusate administered over 90 minutes. The starting dose of Oxaliplatin is 175 mg/m2.
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Starting dose of Oxaliplatin is 175 mg/m2 delivered by hyperthermic intraperitoneal chemotherapy over 90 minutes.
  Other Names: Eloxatin

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of heated intra-abdominal oxaliplatin that can be given to patients with colon cancer. Researchers also want to learn more about the ways that pediatric and young adult colon cancer may be different from colon cancer in adults.

DETAILED DESCRIPTION:
Surgery and Study Drug Administration:

If you are found to be eligible to take part in this study, abdominal surgery will be performed to try to remove as many tumors as possible. The abdominal surgery is not being performed specifically for this research study and would be performed even if you did not take part in this study. You will be given a separate consent form to sign that explains the details and risks of surgery in more detail.

During surgery, the abdomen will be temporarily closed. Then the abdominal wash will begin. During the "abdominal wash," heated oxaliplatin will be delivered through plastic tubing that is connected to a pump into the abdomen. The pump pushes the heated oxaliplatin into the abdomen and then pulls it out and recirculates the oxaliplatin. The skin of the abdomen is temporarily closed during the abdominal wash. The surgeon will also "wash" over the closed area of the surgical site. A pump will be used to pump heated oxaliplatin in and out of the abdomen over 90 minutes while the surgeon gently presses on the abdominal wall so the oxaliplatin reaches all areas in the abdomen. After 90 minutes, the oxaliplatin is removed and the abdomen will be "washed" with saline and all fluid will be removed before the surgeon permanently closes the abdomen with 3 layers of stitches.

Two (2) pea-sized tissue samples (tumor and normal abdominal tissue), 2 tablespoons of blood will be sent to the laboratory of Dr. Scott Kopetz for tissue evaluation and extraction of RNA (genetic material). One (1) tumor sample will be removed before the procedure and the other sample will be removed at the end of the procedure. The samples will be examined under a microscope and DNA (the genetic material in cells) will be removed to look for any changes to the DNA. The results of these tests will not be shared with you, nor will they be used for any decisions regarding your treatment.

There is a chance that the surgeon may decide during the surgery that the abdominal wash will not be performed, for example if the disease has spread to or attached to certain organs. If this occurs, your doctor will discuss other treatment options with you.

Study Visits:

On Day 1 after surgery:

* Blood (about 1 teaspoon) will be drawn for routine tests.
* You will have a physical exam.

On Days 2-5, 11, 14, and 30 after surgery:

* Blood (about 1-3 teaspoons) will be drawn for routine tests.
* You will have a physical exam.
* On Day 30 only, you will have a hearing test.

If the doctor thinks it is needed, you will also have follow up visits at 3 and 6 months after surgery. If these visits occur here at MD Anderson, you will not have a hearing test, but you will have an MRI, CT, or PET-CT scan to check the status of the disease. The 3 and 6 month visits following surgery may be performed at your local doctor's office and/or laboratory.

Length of Study:

You will remain on study for up to 6 months. You will be taken off study if the disease gets worse.

If the study doctor learns that the disease has come back or gotten worse at the 6 month follow-up visit, you may be eligible for a re-perfusion, which is a repeat of the surgery and study drug administration. If you are eligible for a re-perfusion, your participation on this study will end and you will be given a new consent form to sign in order to be re-enrolled back onto this study.

This is an investigational study. Oxaliplatin is FDA approved and commercially available for the treatment of advanced bladder cancer, metastatic testicular cancer, metastatic ovarian cancer, hepatoblastoma, neuroblastoma, metastatic appendiceal cancer, and abdominal mesothelioma. The use of heated oxaliplatin given intra-abdominally in pediatric patients with colon cancer is investigational. The study doctor can explain how the study drug is designed to work.

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9-21 years.
2. Histologically proven colon carcinoma with serosal invasion or peritoneal disease or a history of tumor rupture, and/or ascites
3. Radiologic workup must demonstrate that the disease is confined to the abdominal cavity and/or is controlled outside of the abdominal cavity.
4. Radiologic workup or prior abdominal exploration must be consistent with disease which can be debulked to a residual size of less than or equal to 1 cm thickness
5. Patients must have a minimum expected duration of survival of greater than 6 weeks as determined and documented by the attending surgeon or medical oncologist
6. Patients must not have any systemic illness which precludes them from being an operative candidate as determined by anesthesia preoperative evaluation. This includes but is not limited to, sepsis, liver failure, pregnant or lactating females.
7. Patients must have fully intact mental status and normal neurologic abilities. Intact mental status is defined by 'the capacity to identify and recall one's identity and place in time and space. Assessment of mental status and documentation of fully intact mental status will be completed using physical and mental exam by the referring doctor or oncologist.
8. Patients must have Adequate Renal Function Defined as: Creatinine clearance or radioisotope GFR >/=70ml/min/1.73 m^2 or a serum creatinine based on age/gender less than listed value in the table below: 1 to < 2 years 0.6 mg/dL for both males and females, 2 to < 6 years 0.8 mg/dL for both males and females, 6 to < 10 years 1 mg/dL for both males and females, 10 to < 13 years 1.2 mg/dL for both males and females, 13 to < 16 years 1.5 mg/dL for males and 1.4 mg/dL for females, >/= 16 years 1.7 for males and 1.4 for females
9. Patients will be eligible if the WBC is >/=2000/µl or ANC is >/=1,500 and platelets are >/= 100,000/mm3
10. Patients will be eligible if serum total bilirubin and liver enzymes are </= 2 times the upper limit of normal
11. Patients must be recovered from any toxicity from all prior chemotherapy, immunotherapy, or radiotherapy and be at least 14 days past the date of their last treatment

Exclusion Criteria:

1. Patients will be ineligible if they have any concomitant cardiopulmonary disease which would place them at unacceptable risk for a major surgical procedure
2. Patients will be ineligible if they have disease outside of the abdominal cavity which is uncontrolled
3. Patients will be ineligible if they have a baseline neurologic toxicity of Grade 3 or greater (because of the potential neurotoxicity associated with platinum)
4. Patients who have failed previous intraperitoneal platinum therapy will be ineligible ("Failed" is having disease recurrence </= 3 months.)

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerate Dose (MTD) of Oxaliplatin in Hyperthermic Intraperitoneal Chemotherapy | 3 months
  MTD is highest dose in which 1 or fewer patients in 6 treated experience a dose limiting toxicity (DLT). DLT may occur at any time during the initial hospitalization before discharge following the hyperthermic intraperitoneal chemotherapy (HITC). DLT defined in two ways: Hematologic DLT defined as Grade IV neutropenia, anemia, or thrombocytopenia; and Non-hematologic DLT is any Grade III or IV non-hematologic toxicity excluding Grade III nausea or vomiting, Grade III hepatic toxicity which returns to Grade I within two weeks of the HITC, or before hospital discharge, or Grade III fever occurring after the HITC.

SECONDARY OUTCOMES:
Differences in Genetic Aberrations in Pediatric Colon Cancer Patients and Adult Patients | 6 months
  Descriptive statistics on genetic aberrations provided, either by tabulations of frequencies or summary statistics including numbers, mean, standard deviation, median, minimum and maximum, when appropriate.

OTHER OUTCOMES:
Time to Recurrence After HIPEC in Pediatric, Adolescent and Young Adult Age Colon Cancer Patients | 6 months
  Time to recurrence defined as time from treatment to recurrence (event) or to last follow-up date (censored), using the Kaplan-Meier method, with 95% confidence interval. Evaluation of measurable disease by CT or MRI and physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hayes-Jordan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org